CLINICAL TRIAL: NCT01348295
Title: Pediatric Ventilatory Care in Finland 2010
Status: Completed | Type: Observational
Sponsor: University of Oulu (Other)
Responsible Party: Outi Peltoniemi, Univerisity of Oulu
Other Study IDs: FIN2010
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Mechanical Ventilation; Children; Neonates; Pediatric Intensive Care
Keywords: Mechanical ventilation; Children; Neonates; Pediatric intensive care
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mechanically ventilated children: All children under 16 years of age who are needing mechanical ventilation for any reason.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No interventions are made. The purpose of the study is to find out current practices used in pediatric mechanical ventilation.

SUMMARY:
This observational study includes questionnaires send to doctors in all units treating pediatric patients with mechanical ventilation in Finland. Additionally all units treating pediatric patients with mechanical ventilation are invited to perform a quality control-like follow up for 3 months. Patient identity data is not collected, and no interventions to treatment are made.

ELIGIBILITY:
Inclusion Criteria:

* Age under 16 years
* Mechanical ventilation during the follow up period

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children under 16 years needing mechanical ventilation in Finland from 13th of September 2010 to 19th of December 2010.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The duration of mechanical ventilation | 1-2000 hours
  Compare the duration of mechanical ventilation in different units in Finland

SECONDARY OUTCOMES:
Ventilator parameters | 1-2000hours
  Comparison of ventilator parameters used during mechanical ventilation of children in pediatric-, neonatal- and adult intensive care units.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Oulu, Oulu, North Ostrobothnia, Finland